CLINICAL TRIAL: NCT03391414
Title: Effects of Inhaled Bicarbonate on Airway pH in Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joseph Pilewski (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor-Investigator, Joseph Pilewski, Associate Professor of Medicine and Pediatrics, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PRO09120363
Record Dates: First submitted 2012-06-20; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Cystic Fibrosis
Keywords: thick mucus; obstructive lung disease
MeSH Terms: conditions — Cystic Fibrosis; Lung Diseases, Obstructive | interventions — Sodium Bicarbonate; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- hypertonic bicarbonate (Experimental): subjects will be administered a solution of 8.4% hypertonic bicarbonate by nebulizer
  Interventions: Drug: hypertonic bicarbonate
- hypertonic saline (Active Comparator): subjects will be administered a solution of 7% sodium chloride by nebulizer
  Interventions: Drug: sodium chloride

INTERVENTIONS:
Drug: hypertonic bicarbonate — 8.4% sodium bicarbonate inhaled
  Other Names: sodium bicarbonate
  Arms: hypertonic bicarbonate
Drug: sodium chloride — 7% sodium chloride inhaled
  Other Names: hyper-sal
  Arms: hypertonic saline

SUMMARY:
This study will compare the use of inhaled concentrated sodium chloride solution to an inhaled solution of sodium bicarbonate in an attempt to decrease the thickness and stickiness of the mucus in the lungs of a person with cystic fibrosis. Also, this study is also looking at whether or not it is possible to decrease the acidity of the airways by inhaling sodium bicarbonate through nebulizer treatments.

DETAILED DESCRIPTION:
This study will compare the use of inhaled concentrated sodium chloride solution to an inhaled solution of sodium bicarbonate in an attempt to decrease the thickness and stickiness of the mucus in the lungs of a person with cystic fibrosis. Also, this study is also looking at whether or not it is possible to decrease the acidity of the airways by inhaling sodium bicarbonate through nebulizer treatments.

ELIGIBILITY:
Inclusion Criteria:

1. FEV1 greater than 50% predicted.
2. Ability to spontaneously expectorate sputum (with or without chest physiotherapy).
3. Stable disease as defined by absence of exclusion criteria numbers 3-5 and clinician assessment.

Exclusion Criteria:

1. Reactive airway disease
2. Use of inhaled hypertonic saline in the past 28 days
3. Use of IV antibiotics in the past 4 weeks
4. Changes in CF-related medications in the four weeks prior to study screening
5. SpO2 < 94% on room air or use of supplemental oxygen.
6. Presence of untreated gastroesophageal reflux disease (GERD) or residual acid reflux symptoms in cases of treated GERD more than three times per week.
7. Pregnant or nursing females.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Exhaled breath condensate pH change | two time points (baseline and four (4) hours)
  Change in pH after inhalation of two doses on one day

SECONDARY OUTCOMES:
Expectorated sputum change | two time points (Baseline and four (4) hours)
  Change in sputum wet-to-dry ratio ratio after inhalation of two doses on one day
Spirometry | two time points (baseline and four (4) hours)
  FEV1 before and after inhalation of two doses on one day

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M PIlewski, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Fallk Clinic, Pittsburgh, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No